CLINICAL TRIAL: NCT05330637
Title: Study on the Influence of Climatic and Environmental Factors on Respiratory or Allergic Diseases in Sanya, Hainan Province, China.
Brief Title: Study on the Influence of Climatic and Environmental Factors on Respiratory Diseases in Sanya, Hainan Province, China.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: SYFYIRB2022009
Record Dates: First submitted 2022-03-18; First posted 2022-04-15 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Asthma; Allergic Rhinitis; Chronic Obstructive Pulmonary Disease(COPD); Atopic Dermatitis; Eczema; Urticaria; Bronchitis; Bronchiectasis Adult; Emphysema
Keywords: Asthma; Allergic Rhinitis; Climatotherapy; Chronic Obstructive Pulmonary Disease(COPD); Atopic Dermatitis; Climate; Environment
MeSH Terms: conditions — Asthma; Rhinitis, Allergic; Pulmonary Disease, Chronic Obstructive; Dermatitis, Atopic; Eczema; Urticaria; Bronchitis; Emphysema | interventions — Climate; Environment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Veinal blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- Migratory old people with asthma from northern China in Sanya: Migratory old people with asthma from northern China to Sanya have being exposure to two different climate and environment from northern China to Sanya for months.
  Interventions: Other: Climate and environment in Sanya
- Migratory old people with allergic rhinitis from northern China in Sanya: Migratory old people with allergic rhinitis from northern China to Sanya have being exposure to two different climate and environment from northern China to Sanya for months.
  Interventions: Other: Climate and environment in Sanya
- Migratory old people with Chronic Obstructive Pulmonary Disease (COPD) from northern China in Sanya: Migratory old people with Chronic Obstructive Pulmonary Disease (COPD) from northern China to Sanya have being exposure to two different climate and environment from northern China to Sanya for months.
  Interventions: Other: Climate and environment in Sanya
- Migratory old people with atopic dermatitis from northern China in Sanya: Migratory old people with atopic dermatitis from northern China to Sanya have being exposure to two different climate and environment from northern China to Sanya for months.
  Interventions: Other: Climate and environment in Sanya
- Children with asthma in Sanya: Children with asthma have being exposure to tropical climate and environment in Sanya for years.
  Interventions: Other: Climate and environment in Sanya
- Children with allergic rhinitis in Sanya: Children with allergic rhinitis have being exposure to tropical climate and environment in Sanya for years.
  Interventions: Other: Climate and environment in Sanya
- Children with atopic dermatitis in Sanya: Children with atopic dermatitis have being exposure to tropical climate and environment in Sanya for years.
  Interventions: Other: Climate and environment in Sanya
- Children with eczema in Sanya: Children with eczema have being exposure to tropical climate and environment in Sanya for years.
  Interventions: Other: Climate and environment in Sanya
- Children with urticaria in Sanya: Children with urticaria have being exposure to tropical climate and environment in Sanya for years.
  Interventions: Other: Climate and environment in Sanya
- Migratory old people with eczema from northern China in Sanya: Migratory old people with eczema from northern China to Sanya have being exposure to two different climate and environment from northern China to Sanya for months.
  Interventions: Other: Climate and environment in Sanya
- Migratory old people with urticaria from northern China in Sanya: Migratory old people with urticaria from northern China to Sanya have being exposure to two different climate and environment from northern China to Sanya for months.
  Interventions: Other: Climate and environment in Sanya

INTERVENTIONS:
Other: Climate and environment in Sanya — Sanya have unique island climate and environment campared with the north of China, with a feature of warm, moist and long-sunshine.

SUMMARY:
To investigate the Influence of Climatic and Environmental Factors on Respiratory or Allergic Diseases in Sanya.

DETAILED DESCRIPTION:
The study is an observational research, which will recruit the community migratory old people and children at school using cluster sampling in Sanya by Sanya Maternal and Child Health Care Hospital (Sanya Women and Children's Hospital). Sanya Central Hospital(Hainan Third People's Hospital) and People's Hospital of Sanya will assist to diagnose old people disease. The data of climate and environment will be obtained from Sanya Meteorological Administration and Sanya Municipal Ecology and Environment Bureau.

1. The primary purpose is to investigate the influence of the unique tropical climate and environmental factors on the migratory old people with diseases such as asthma, allergic rhinitis, COPD or atopic dermatitis in Sanya from northern China, and to provide scientific evidence for publicity of the tourism and the health care industry.
2. The secondary purpose is to investigate prevalence and risk factors of asthma, allergic rhinitis and atopic dermatitis among children in Sanya, which will provide a base for prevention and control strategies.
3. The third purpose is to retrospectively analyze the influence of climate and environmental factors in Sanya on children with asthma, allergic rhinitis and atopic dermatitis in the past decade, and a comparative analysis of the incidence on children in Sanya and Shanghai.

ELIGIBILITY:
Inclusion Criteria:

* 50-80 years-old migratory people with asthma, allergic rhinitis, COPD or atopic dermatitis from northern China;
* 3-12 years-old children in Sanya;
* Agree to participate this study.

Exclusion Criteria:

* Disagree to participate this study;
* Having other respiratory diseases which can influence airflow, such as lung cancer, tuberculosis, pneumonia, bronchiectasis, etc;
* Inability to understand the study procedures or inability/reluctance to answer questionnaire judged by the investigator.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. 50-80 years-old migratory people with asthma, allergic rhinitis, COPD or atypical dermatitis from northeast China.
  2. 3-12 years-old children with asthma, allergic rhinitis, atypical dermatitisin in Sanya.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
The difference of migratory old people with asthma, COPD, allergic rhinitis or atopic dermatitis between winter-spring season in tropical Sanya, Hainan Island and summer-autumn season in northeast China. | 3 year
  The asthma, COPD, allergic rhinitis or atopic dermatitis will be diagnosed and assessed through history of diseases and questionnaire..

SECONDARY OUTCOMES:
Asthma control of migratory old people with asthma. | 1-3 year
  Quality of life is assessed through questionnaires of "Asthma Control Questionnaire (ACQ) ".
Asthma life quality of migratory old people with asthma. | 1-3 year
  Quality of life is assessed through questionnaires of "Asthma Quality of Life Questionnaire (AQLQ)".
Lung function of migratory old people with asthma or COPD. | 1-3 year
  Lung function is assessed through simple lung function test using spirometry.
The respiratory function of migratory old people with COPD. | 1-3 year
  Lung function is assessed through Saint George Respiratory Questionnaire (SGRQ).
Allergens will be detected in migratory old people with asthma, allergic rhinitis or atopic dermatitis. | 1-3 year
  Veinal blood was extracted to detect allergens.
Inflammatory factors will be detected in migratory old people with asthma, allergic rhinitis or atopic dermatitis. | 1-3 year
  Inflammatory factors such as esophageal granulocytes and eosinophils will be detected to assess inflammatory status of the migratory old people.
The change of asthma incidence rate in migratory old people . | 1-3 year
  Diagnosis and severity grading of asthma is based on the "American Thoracic Society" or the "National Heart, Lung, and Blood Institute guidelines."

CONTACTS AND LOCATIONS:
Overall Officials: Shijian Liu, Ph.D, Principal Investigator — Shanghai Children's Medicial Center affiliated Shanghai Jiao Tong University School of Medicine
Locations (1):
- Sanya Women and Children's Hospital, Shanghai Children's Medical Center, School of Medicine, Shanghai Jiao Tong University, Sanya, Hainan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang K, Yang T, Xu J, Yang L, Zhao J, Zhang X, Bai C, Kang J, Ran P, Shen H, Wen F, Chen Y, Sun T, Shan G, Lin Y, Xu G, Wu S, Wang C, Wang R, Shi Z, Xu Y, Ye X, Song Y, Wang Q, Zhou Y, Li W, Ding L, Wan C, Yao W, Guo Y, Xiao F, Lu Y, Peng X, Zhang B, Xiao D, Wang Z, Chen Z, Bu X, Zhang H, Zhang X, An L, Zhang S, Zhu J, Cao Z, Zhan Q, Yang Y, Liang L, Tong X, Dai H, Cao B, Wu T, Chung KF, He J, Wang C; China Pulmonary Health (CPH) Study Group. Prevalence, risk factors, and management of asthma in China: a national cross-sectional study. Lancet. 2019 Aug 3;394(10196):407-418. doi: 10.1016/S0140-6736(19)31147-X. Epub 2019 Jun 20. PMID 31230828
- [Result] Xie L, Liu Z, Hao S, Wu Q, Sun L, Luo H, Yu R, Li X, Wu X, Li S. Assessment of knowledge, attitude, and practice towards pulmonary rehabilitation among COPD patients: A multicenter and cross-sectional survey in China. Respir Med. 2020 Nov-Dec;174:106198. doi: 10.1016/j.rmed.2020.106198. Epub 2020 Oct 20. PMID 33120194
- [Result] Zhu B, Wang Y, Ming J, Chen W, Zhang L. Disease burden of COPD in China: a systematic review. Int J Chron Obstruct Pulmon Dis. 2018 Apr 27;13:1353-1364. doi: 10.2147/COPD.S161555. eCollection 2018. PMID 29731623
- [Result] Ding Y, Xu J, Yao J, Chen Y, He P, Ouyang Y, Niu H, Tian Z, Sun P. The analyses of risk factors for COPD in the Li ethnic group in Hainan, People's Republic of China. Int J Chron Obstruct Pulmon Dis. 2015 Nov 30;10:2593-600. doi: 10.2147/COPD.S86402. eCollection 2015. PMID 26664107
- [Result] Garcia-Almaraz R, Reyes-Noriega N, Del-Rio-Navarro BE, Berber A, Navarrete-Rodriguez EM, Ellwood P, Garcia Marcos Alvarez L; GAN Phase I group. Prevalence and risk factors associated with allergic rhinitis in Mexican school children: Global Asthma Network Phase I. World Allergy Organ J. 2020 Dec 5;14(1):100492. doi: 10.1016/j.waojou.2020.100492. eCollection 2021 Jan. PMID 34659624
- [Result] Pesce G, Bugiani M, Marcon A, Marchetti P, Carosso A, Accordini S, Antonicelli L, Cogliani E, Pirina P, Pocetta G, Spinelli F, Villani S, de Marco R. Geo-climatic heterogeneity in self-reported asthma, allergic rhinitis and chronic bronchitis in Italy. Sci Total Environ. 2016 Feb 15;544:645-52. doi: 10.1016/j.scitotenv.2015.12.015. Epub 2015 Dec 10. PMID 26674694
- [Result] Zanolin ME, Pattaro C, Corsico A, Bugiani M, Carrozzi L, Casali L, Dallari R, Ferrari M, Marinoni A, Migliore E, Olivieri M, Pirina P, Verlato G, Villani S, Marco R; ISAYA Study Group. The role of climate on the geographic variability of asthma, allergic rhinitis and respiratory symptoms: results from the Italian study of asthma in young adults. Allergy. 2004 Mar;59(3):306-14. doi: 10.1046/j.1398-9995.2003.00391.x. PMID 14982513
- [Result] Weiland SK, Husing A, Strachan DP, Rzehak P, Pearce N; ISAAC Phase One Study Group. Climate and the prevalence of symptoms of asthma, allergic rhinitis, and atopic eczema in children. Occup Environ Med. 2004 Jul;61(7):609-15. doi: 10.1136/oem.2002.006809. PMID 15208377
- [Result] Wang X, Zhuang Y, Chen Y, Wang H, Wang X. Prevalence of adult eczema, hay fever, and asthma, and associated risk factors: a population-based study in the northern Grassland of China. Allergy Asthma Clin Immunol. 2021 Mar 9;17(1):27. doi: 10.1186/s13223-021-00532-7. PMID 33750462
- [Result] Su N, Lin J, Chen P, Li J, Wu C, Yin K, Liu C, Chen Y, Zhou X, Yuan Y, Huang X. Evaluation of asthma control and patient's perception of asthma: findings and analysis of a nationwide questionnaire-based survey in China. J Asthma. 2013 Oct;50(8):861-70. doi: 10.3109/02770903.2013.808346. PMID 23713625
- [Result] Li J, Sun B, Huang Y, Lin X, Zhao D, Tan G, Wu J, Zhao H, Cao L, Zhong N; China Alliance of Research on Respiratory Allergic Disease. A multicentre study assessing the prevalence of sensitizations in patients with asthma and/or rhinitis in China. Allergy. 2009 Jul;64(7):1083-92. doi: 10.1111/j.1398-9995.2009.01967.x. Epub 2009 Feb 11. PMID 19210346
- [Result] Donaldson GC, Wedzicha JA. The causes and consequences of seasonal variation in COPD exacerbations. Int J Chron Obstruct Pulmon Dis. 2014 Oct 6;9:1101-10. doi: 10.2147/COPD.S54475. eCollection 2014. PMID 25336941
- [Result] Kantor R, Silverberg JI. Environmental risk factors and their role in the management of atopic dermatitis. Expert Rev Clin Immunol. 2017 Jan;13(1):15-26. doi: 10.1080/1744666X.2016.1212660. Epub 2016 Jul 28. PMID 27417220
- [Result] Wang X, Li LF, Zhao DY, Shen YW. Prevalence and Clinical Features of Atopic Dermatitis in China. Biomed Res Int. 2016;2016:2568301. doi: 10.1155/2016/2568301. Epub 2016 Nov 13. PMID 27957490